CLINICAL TRIAL: NCT00930306
Title: A Phase I, Open Label, Multi Centre Study in Healthy Volunteers to Estimate the Effect of Multiple Doses of AZD2066 on the Activity of CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6 and CYP3A4 by Administering a Cocktail of Caffeine, Bupropion, Tolbutamide, Omeprazole, Metoprolol and Midazolam
Brief Title: AZD2066 Cocktail Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D0475C00011
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; AZD2066
MeSH Terms: conditions — Chronic Pain | interventions — AZD2066; Caffeine; Tolbutamide; Drugs, Generic; Omeprazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 12 AZD2066 Capsule, 2 mg & 8 mg 2 Caffeine Tablet, 2 x 50 mg 2 Tolbutamide Tablet, half of 500 mg 2 Omeprazole Tablet, 20 mg 2 Midazolam Tablet, 7.5 mg 2 Metoprolol Tablet, 100 mg 2 Bupropion Tablet, 150 mg
  Interventions: Drug: AZD2066; Drug: Caffeine; Drug: Tolbutamide; Drug: Omeprazole Tablet, 20 mg; Drug: Midazolam Tablet, 7.5 mg

INTERVENTIONS:
Drug: AZD2066 — 12 doses, Given as capsule, 2 mg & 8 mg
Drug: Caffeine — 2 doses, Given as Tablet, 2x50 mg
  Other Names: Pharmapac/ProPlus®
Drug: Tolbutamide — 2 doses, Given as Tablet, half of 500 mg
  Other Names: Actavis /generic
Drug: Omeprazole Tablet, 20 mg — 2 doses, Given as Tablet, 20 mg
  Other Names: AstraZeneca/Losec® MUPS®
Drug: Midazolam Tablet, 7.5 mg — 2 doses, Given as Tablet, 7.5 mg
  Other Names: Roche/generic

SUMMARY:
The aims of this study are to examine the effect of repeated doses of AZD2066 and of caffeine, bupropion, tolbutamide, omeprazole, metoprolol and midazolam on the blood concentrations of each other

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Healthy volunteers with BMI between 18 and 30 kg/m2
* Medical and surgical history and physical examination without any clinically significant findings
* Non smokers or past smokers who have stopped smoking within the last 6 months.

Exclusion Criteria:

* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, personality disorder or other significant psychiatric disorders or any other major disorder that may interfere with the objectives of the study, as judged by the Investigator
* Clinically significant illness as judged by the Investigator, within four weeks before the first administration of investigational product.
* Female subjects who have a positive pregnancy test or who are pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | Frequent sampling occasions during

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Lilja, Study Director — AstraZeneca R&D, Södertälje, Sweden; Simon Constable, Principal Investigator — ICON Development Solutions, Manchester, UK
Locations (2):
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester